CLINICAL TRIAL: NCT06238414
Title: Attempted Suicide Intervention Treatment and Prevention: a Randomised Controlled Trial
Brief Title: Attempted Suicide Intervention Treatment and Prevention (SAMIT Program)
Acronym: SAMIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)463/2022
Record Dates: First submitted 2023-11-20; First posted 2024-02-02 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Suicide, Attempted; Suicide Prevention
Keywords: Medically serious suicide attempts (MSSA); Psychotherapy; Intervention; Randomized controlled trial
MeSH Terms: conditions — Suicide, Attempted; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: An experimental, randomized controlled trial will be conducted with patients hospitalized after a MSSA. The case group will receive an 8-session early psychological intervention while the control group will be treated as usual. The intervention consists of eight face-to-face sessions that include techniques from the narrative theory, dialectical behavioral (DBT), mentalization-based therapy orientation (MBT) and narrative approach, concretely an adaptation from the ASSIP therapy. Longitudinal assessment will be conducted at baseline and 3, 6 and 12 months after the early psychological intervention. The main outcome will be re-attempting suicide during the follow-up period. Secondary outcomes measures will be related to: biological (biomarkers), psychosocial (quality of life and reasons for living) and clinical (psychometric assessments, psychopathological status and suicidiological variables) factors.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/case participant (Experimental): The case group will receive an 8-session early psychological intervention
  Interventions: Other: Early psychotherapeutic intervention
- Control case/participant (No Intervention): The control group will be treated as usual (TAU)

INTERVENTIONS:
Other: Early psychotherapeutic intervention — The case group will receive an 8-session early psychological intervention The intervention consists of eight face-to-face sessions that include techniques from the dialectical behavioral (DBT), mentalization based therapy orientation (MBT), and narrative approach, concretely an adaptation from the ASSIP therapy. The sessions will be conducted by a clinical psychologist with expertise in psychotherapy. There will be two 60-minutes sessions per week.
  Arms: Intervention/case participant

SUMMARY:
Suicide has become a first-order public health concern after the negative impact of coronavirus disease 2019 (COVID-19) on the mental health of the general population. Few studies have analyzed the effects of early psychotherapeutic interventions on subjects who have attempted suicide, and even fewer focus on those hospitalized in nonpsychiatric units after a medically serious suicide attempt (MSSA). The most important risk factor for attempting suicide is having made a previous suicide attempt. Subjects are also at higher risk the first year after the attempt.

The main aim of this study is to evaluate the effectiveness of individual psychological treatment with patients hospitalized after a MSSA. The secondary objectives are: 1) acknowledge the evolution of the incidence of MSSA hospitalized during the pandemic; 2) analyze the impact of the psychological intervention using biological, psychosocial, and clinical variables. An experimental, controlled, and randomized trial will be conducted with patients older than 16 admitted to two general hospitals. The case group will receive an 8- session of individual psychotherapy while the control group received treatment as usual. Longitudinal assessment will be conducted at baseline, post-treatment, and 3, 6, and 12 months after.

The main outcome variable will be re-attempting suicide during the follow-up.

DETAILED DESCRIPTION:
In the last decades, many studies have tried to analyse the risk and protective factors related to suicidal behaviors. However, there are fewer studies evaluating the effectiveness of early psychotherapeutic interventions with subjects who have attempted suicide, and even fewer based on subjects who have been hospitalised after a medically serious suicide attempt (MSSA). This type of attempt can be considered a nearly lethal suicide attempt, and it usually has serious medical and psychological consequences. On the other hand, having a previous suicide attempt is known to be the most important risk factor for a subsequent attempt. Moreover, the first year after the attempts is the highest-risk period to re-attempt.

The main objective of this study is to evaluate the effectiveness of an early individual psychotherapeutic intervention with subjects hospitalised after a MSSA. The secondary objectives are: 1) to study how the incidence of MSSA needing hospitalisation has evolved during the pandemic; and 2) to study the impact of the psychotherapeutic intervention on several biological, psychosocial, and clinical variables.

This study is expected reducing the risk of re-attempting suicide and improving their quality of life and wellbeing. It may also provide valuable insight with regards to the relationship between this improvement and some correlated biological and psychosocial changes.

A randomised, controlled trial will be conducted with patients at 2 general hospitals in Catalonia (Hospital Vall d'Hebron and Hospital Clinic) after a MSSA. The case-intervention group will receive an 8-session early individual psychotherapy and the control group will receive the treatment-as-usual intervention (TAU). The intervention consists of eight face-to-face sessions that include techniques from dialectical-behavioural (DBT), cognitive-behavioural (CBT), mentalization treatment (MBT), and narrative approaches, based on an adaptation of the Attempted Suicide Short Intervention Program (ASSIP). The sessions will be conducted by a psychologist with expertise in psychotherapy. There will be two 60-minute sessions per week.

The subjects will be periodically assessed at baseline (before the treatment) and post-treatment. We also monitored during the follow-up period, at 3, 6, and 12 months after the end of the treatment.

In order to ascertain the effects of the psychotherapeutic intervention, several types of variables will be studied: biological (blood inflammatory biomarkers), psychosocial (quality of life, reasons for living, and personality dimensions), and clinical (related to the psychopathological status and to suicidal behaviors). The incidence of patients needing hospitalisation after a MSSA during the pandemic will also be analysed.

Socio-demographic variables will also collected during the baseline assessment. It will include information on: age; sex; nationality; civil status; educational level; employment status; family situation; history of child/adolescent/adult trauma or abuse; history of personal medical or surgical conditions; and current medical or surgical conditions.

Blood samples will be drawn before and after treatment, by an experienced nurse between 7.00 and 10.00 a.m. of the scheduled day after an overnight fasting. Laboratory analyses will be conducted on the same day as the clinical assessments.Complete and differential white blood cell (WBC) count (by an automated analyzer) acute-phase reactants (i.e., high-sensitivity C-reactive protein (hsCRP)) (by an automated analyzer) - Pro-inflammatory cytokines [Interleukine 6 (IL-6)]. Lipid profile (i.e., cholesterol, LDL, HDL, very low density lipoprotein (VLDL), triglycerides, Poly-Unsaturated Fatty Acids (PUFA's) (by an automated analyzer). In addition, serum and/or plasma will be separated by centrifugation, aliquoted, and immediately placed at -80°C until the time of analysis of the following metabolites: Tryptophan and Kynurenine pathway metabolites (i.e., Tryptophan (TRP), serotonin (5-HT), Kynurenine (KYN), kynurenic acid (KYNA), Xanthurenic acid (XA), 3-hydroxykynurenine (3-HK), 3-hydroxyanthranilic acid (3-HAA), Quinolinic acid (QUIN), Picolinic acid (PIC) by liquid chromatography-tandem mass spectrometry (LCMS/MS). Blood samples will be obtained at each hospital and kept frozen at -80 °C. Once the study is completed, the Clinic Hospital samples will be sent to the University Vall d'Hebron Hospital laboratory for analysis, along with all other samples.

ELIGIBILITY:
Inclusion Criteria:

* Older than 16 years.
* Remaining hospitalized for 24 hours or more at HUVH and HCP after a MSSA for 24 or more (> = 24 hours).
* Needing specialized care units (including Intensive Care Units, Hyperbaric Camera Units, Burned Units, Semicritical Units)
* Needing specialized surgical treatment, excluding superficial cuts
* Needing extensive medical treatment and observation (gastric lavage, activated charcoal, observation of neurological tests or other complementary tests)
* MSSA with high lethality methods (precipitation, hanging, firearm, stabbing) needing hospitalization for 24 or more hours, regardless of the treatment unit.

Exclusion Criteria:

* Patients with suicide attempts who were discharged in <24 h
* Patients under 16 years.
* Patients with mild to severe cognitive impairment.
* Lack of informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Number of suicide attempts (recurrence) | 1 year
  The recurrence of the suicide attempt will be monitored by two mechanisms:
  1. During follow-up evaluations at 3, 6, and 12 months through a telephone call to the patient
  2. Reviewing the patient's medical history through the hospital's public health system program.
  The variable will be recorded by a dicotomic answer: "YES" if the patient had an intent during the follow-up period (3, 6, and 12 months) and "NO" if the patient did not have an intent. In cases of reattempt, the C-SSRS, SCS, and SALSA scales will be administered. In case of consummated attempts, information will be collected through clinical history and family interviews if it's required.
  We expected that the "case-intervention group" would have fewer re-attempts than the control group.
Severity of suicide behaviour | 1 year
  The investigators will evaluate the suicide severity through the C-SSRS scale in the pre-treatment phase only if the patient makes a suicide attempt or has a suicide ideation during the study pre and post-treatment and follow up perios (3,6 and 12 months) .
  Columbia Suicide Severity Rating Scale (C-SSRS) is a semi-structured interview with dicothomic answers (yes or no) that captures the occurrence, severity, and frequency of suicide-related behaviour and thoughts during the assessment period.
Suicide behaivour | 1 year
  The investigators evaluated the suicide attempt trought the SCS scale in pre treatment phase and only if the patient makes a suicide attempt or has a suicide ideation during the study pre and post-treatment and follow up perios (3,6 and 12 months) .
  Suicidal Crisis Syndrome (SCS): This is an interview with dichotomous responses that assess conditions linked to imminent suicidal behavior characterized by (a) affective disturbance, loss of cognitive control, hyperarousal and social withdrawal (Criterion B) and (b) a generalized sense of entrapment in which leaving an intolerable life situation is perceived as both urgent and impossible.
Lethality of suicide attempt | 1 year
  In the baseline phase, before treatment, we assess the lethality of the suicide attempt through the Scale for Assessment of the Lethality of the Suicide Attempt (SALSA). The investigators will only administer the scale again in case of re-attempt during the follow-up.
  SALSA consists of two parts: The first component has four items indicating seriousness of the attempt and its likely consequences and the second component is the global impression of lethality. All the items are scored from 1 to 5, higher scores suggestive of increased lethality

SECONDARY OUTCOMES:
Well-being: Intrapsychic functions, Interpersonal relationships, Instrumental role, Use of common objects and daily activities. | 1 year
  After psychotherapeutic intervention, the investigators expected to improve the well-being of the patients. We compared between pre- and post-treatment. This variable will be mesured through the Quality of life test (QoL) in the follow-up (3, 6, and 12 months).It consists of 21 items that are grouped into the following 4 categories or factors: Intrapsychic functions: cognition, cognition and affectivity (items 13-17, 20-21).Interpersonal relationships: interpersonal and social experience (items 1-8).Instrumental role: work, study, parental duties (items 9-11).Use of common objects and daily activities (items 18-19).Item 12 (satisfaction) does not score in any of the factors. Each item is scored according to a 7-value Likert scale, ranging from 0 (highest degree of dysfunction in that item) to 6 (normal). The time frame of reference is the previous 4 weeks.
  The higher the score, the higher the quality of life in each dimension.
Psychological Pain | 1 year
  After psychotherapeutic intervention, the investigators expected to improve the psychological pain of the patients. This variable will be compared between pre- and post-treatment through the Psychological Pain Scale (PS-E) and will also be assessed in the follow-up (3, 6, and 12 months).
  The scale evaluates psychological pain as a subjective experience. It is composed of 13 items with a Likert-type response format (1-5) from lowest (1) to highest pain score (5).
  The higher scores higher psychological pain.
Anxiety and Depression | 1 year
  After psychotherapeutic intervention, the investigators expected to improve the anxiety and depression symptoms. This variable will be compared between pre- and post-treatment and also assessed through the Hospital Anxiety and Depression Scale (HADS) in the follow-up (3, 6, and 12 months).
  Anxiety and Depression Scale (HADS) : consists in 14 items on a 4-point Likert scale (range 0-3) with three denoting highest anxiety or depression level. Its seven items for each subscale (anxiety and depression). The sum of the 14 items makes up the overall score.
Impulsivity | 1 year
  After psychotherapeutic intervention, the investigators expected to decrease the impulsivity of the patients. This variable will be compared between pre- and post-treatment and also assessed through the Barrat Impulsiveness Scale (BIS-11) in the follow-up (3, 6, and 12 months).
  BIS-11 is a widely used 30 question self-report measure of impulsiveness. It includes six first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and three second-order factors (attentional, motor, and non-planning impulsiveness). It is rated on a four-point Likert scale of 1 = Rarely/Never to 4 = Almost Always/Always. The total scores can range from 30 to 120. However, higher scores on the BIS-11 reflect higher levels of impulsiveness.
Interleukin 6 (IL-6) | 1 month
  The change in a set of IL-6 (pg/mL) will be assessed from baseline to the end of the intervention at week 4.
Suicide intentionality | 1 year
  In the baseline phase, before treatment, we assess the suicide intentonality through the Beck suicidal intentionality scale (SIS). The investigators will only administer the scale again in case of re-attempt during the follow-up.
  SIS: is a semi-structured scale consisting of 20 items, which are rated on a 3-point scale (0 to 2 points). Scores can range from 0 to 38, with higher values indicating a greater risk of suicide.
Reflective capacity | 1 year
  After psychotherapeutic intervention, the investigators expected to improve the reflective functioning of the patients. This variable will be compared between pre- and post-treatment and also assessed through the Reflective Functioning Questionnaire (RFQ-8) in the follow-up (3, 6, and 12 months).
  RFQ-8 is a self-administered questionnaire that consists of 8 items. It provides responses for each item on a seven-point scale between "strongly disagree" and "strongly agree" response options. The higher the score, the worse the reflective capacity.
Suicide ideation | 1 year
  After psychotherapeutic intervention,the investigators expected to decrease and/or eliminate the suicide ideation. This variable will be compared between pre- and post-treatment and during follow-up evaluations at 3, 6, and 12 months through the the Scale for Suicide Ideation (SSI).
  SSI evaluates the presence and intensity of suicidal thoughts in a week before evaluation. It is composed of 19 items that are scored from 0 to 2, where 0 corresponds to moderate to strong, 1 to weak, and 2 to no suicide ideation.
Hopelessness | 1 year
  After psychotherapeutic intervention, the investigators expected to improve the anxiety and depression symptoms. This variable will be compared between pre- and post-treatment and also assessed through the Beck Hopelessness Scale (BHS) tests in the follow-up (3, 6, and 12 months).
  Beck Hopelessness Scale (BHS): is a 20-item with true-false test answers. Scores ranging from: 0 to 3 as are considered within the normal range, 4 to 8 identify mild hopelessness, scores from 9 to 14 identify moderate hopelessness, and scores greater than 14 identify severe hopelessness.
C-reactive protein | 1 month
  The change in a set of C-reactive protein (mg/dL) will be assessed from baseline to the end of the intervention at week 4:
White Blood Cells (x10E9/L) | 1 month
  The change in a set of White Blood Cell count (x10E9/L) will be assessed from baseline to the end of the intervention at week 4:
Cholesterol (mg/dL) | 1 month
  The change in a set of Cholesterol, will be assessed from baseline to the end of the intervention at week 4.
High-Density Lipoprotein (HDL) (mg/dL) | 1 month
  The change in a set of HDL (mg/dL) will be assessed from baseline to the end of the intervention at week 4.
Low -Density Lipoprotein (LDL) (mg/dL) | 1 month
  The change in a set of LDL will be assessed from baseline to the end of the intervention at week 4.
Tryglycerides (mg/dL) | 1 month
  The change in a set of tryglycerides will be assessed from baseline to the end of the intervention at week 4.
Attachment | 1 month
  In the pre-treatment phase, the investigators will assess the attachment of the patient with the CAMI-R short version test in order to study the relationship between the type of attachment and suicide behaviour.
  Short version of CaMir questionnaire (CaMir-R)(65)) is a self-questionnaire that measures attachment representations. It is based on the subject's evaluations of past and present attachment experiences and family functioning. It consists of 32 items to be answered by the participant on a 5-point Likert-type scale (1 = strongly disagree, 5 = strongly agree). The questionnaire consists of seven dimensions, five of which refer to attachment representations (security: availability and support of attachment figures; family preoccupation; parental interference; self-sufficiency and resentment against parents; and childhood trauma), and the remaining two refer to representations of family structure (value of parental authority and parental permissiveness).
Cognition | 1 month
  Before starting the treatment, the patient will undergo the Montreal Cognitive Assessment (MOCA) to control for cognitive impairment. MOCA will be administered again in the post-treatment phase.
  The MoCA Test, also known as the Montreal Cognitive Assessment, has been proven to be an extremely sensitive method for identifying moderate cognitive impairment (MCI) in its early stages. The MoCA exam is scored, with a maximum of thirty being possible. It takes ten to twelve minutes to finish. The MoCA test uses a total of 11 distinct exercises and tasks to assess seven domains (aspects) of cognitive function: attention and executive function, language domains, memory, abstraction, calculation, and orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dolores Braquehais, Principal Investigator — VHIR; Pol Bruguera, Principal Investigator — Hospital Clínic-IDIBAPS
Locations (1):
- Anna Beneria, Barcelona, Spain

REFERENCES:
- [Derived] Beneria A, Motger-Alberti A, Quesada-Franco M, Arteaga-Henriquez G, Santesteban-Echarri O, Ibanez P, Parramon-Puig G, Sanz-Correcher P, Galynker I, Ramos-Quiroga JA, Pintor L, Bruguera P, Braquehais MD. A Suicide Attempt Multicomponent Intervention Treatment (SAMIT Program): study protocol for a multicentric randomised controlled trial. BMC Psychiatry. 2024 Oct 8;24(1):666. doi: 10.1186/s12888-024-06113-3. PMID 39379877